CLINICAL TRIAL: NCT05395663
Title: Effectiveness and Scalability of a Home Health Navigator Program to Reduce Environmental Hazards
Brief Title: Scalability of a Home Health Navigator Program to Reduce Arsenic, Nitrate, and Lead in Private Well Water
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: Oregon Health Authority (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Molly Kile, Co-Principal Investigator, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NIH # 5R01ES031669; R01ES031669 (NIH)
Record Dates: First submitted 2022-05-10; First posted 2022-05-27 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Pollution; Exposure
Keywords: drinking water; arsenic; nitrate; lead; environmental pollution; ground water; home environment; water wells; health promotion; water pollutant; water pollution; water treatment; water purification; chemical water pollution; underground water; water quality; environmental carcinogens; environmental health; environmental exposure; environmental pollutant; toxic environmental substances
MeSH Terms: interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The care providers are the OSU Extension Service agents serving as the navigators in the intervention arm and the Oregon Health Authority as the usual care arm. They will not know participants assigned to the other arms. Biostatistician will evaluate the effectiveness of the intervention without knowing the condition of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Usual practice (Active Comparator): People will receive a free well water test kit that is delivered by mail and the results from this water test. They will also be mailed material that is provided by the Oregon Health Authority's Domestic Well Stewardship Program which is the Water Well Owner's Handbook(in English or Spanish) and contaminant guides.
  Interventions: Behavioral: Community health worker
- Arm 2: Health navigator (Experimental): People will receive a free well water test kit that is delivered by mail and the results from this water test. They will also be mailed material that is provided by the Oregon Health Authority's Domestic Well Stewardship Program which is the Water Well Owner's Handbook(in English or Spanish) and contaminant guides. In addition, a trained health navigator will meet with the homeowner three times to assist the homeowner's decision-making.
  Activities include: i) Interpreting results, ii) Improving health literacy and numeracy through teach-back moments, iii) Assessment of household risk for contaminants from well and septic, iv) Assessment of risk to family members, pets, livestock, etc v) Coaching to resolve ambivalence or lack of motivation and other barriers using elicit-provide-elicit motivational interviewing; vi) Assistance with decision-making and weighing financial options, and vii) Goal-setting and action plans.
  Interventions: Behavioral: Community health worker

INTERVENTIONS:
Behavioral: Community health worker — A trained navigator (e.g. OSU Extension staff) will have 3 meetings with the participants in Arm 2. These meetings will be held in person, on the phone, or in zoom.

SUMMARY:
Approximately 34 million Americans rely on private wells to supply their drinking water. Private wells are excluded from the Safe Drinking Water Act. Consequently, people who use private wells have not benefited from pollution prevention activities mandated by this law. This is a public health concern because toxic chemicals such as arsenic, nitrate, and lead are frequently detected in drinking water provided by private wells at concentrations that exceed the Safe Drinking Water Act's maximum contaminant levels. Chronic exposure to toxics in drinking water increase the risk of several chronic diseases. Several states in the U.S. have implemented or are proposing legislative policies to require testing and treatment of private wells and it is critical that public health agencies offer a program to aid homeowners with adherence to these new policies. Subsequently, there is a need to determine if individual-level interventions would be more effective for promoting behaviors that would reduce, mitigate, or eliminate exposure to contaminated well water. Lay health care workers may be able to provide cost-effective counseling to promote environmental health decision making among homeowners that have contaminated wells. This study will involve a community efficacy trial that brings together university-based researchers, State and Local agencies, and Extension Services. The community efficacy trial will be implemented by community health navigators via the Extension service. Specifically, it will involve a randomized controlled trial in Oregon to test the acceptability, fidelity, scalability and efficacy of 2 different intervention arms to reduce harmful toxicant exposures through the adoption of appropriate well water treatment. Upon completion, it will will produce a private well safety intervention program that has been tested and modified through empirical research. By capturing the costs and retaining the most efficacious intervention components, our cooperative approach has a better chance of scalability into practice across multiple stakeholders (i.e. Extension services, state health agencies). This information has the potential to reduce health disparities in rural America that are related to a household's source of drinking water.

ELIGIBILITY:
Participants are eligible for the study if they 1) Reside in Oregon; 2) Are a homeowner with a private well; 3) Use a private well as the primary source of drinking water; 4) Currently live in the home with the private well and intend to live in the home for at least 12 months from now; 5) Be at least 21 years old; and 6) Be able to complete a questionnaire in English or Spanish.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Treatment implemented by homeowner that will reduce their exposure to arsenic, nitrate or lead in their drinking water | 12 months
  The homeowner has adopted behaviors that will be appropriate for reducing their exposure to arsenic, nitrate, and lead in their drinking water. This will be assessed based on the homeowners response on a survey delivered after 12 month. Appropriate treatment will be defined as the use of drinking water technology that removes the contaminant detected (e.g. reverse osmosis, distillation, arsenic removal filter, or removal of lead-based water fixtures) or switching to bottled water for drinking and cooking.
Clean water sample | 12 months
  A water sample that is collected from their home's kitchen faucet is tested by a certified laboratory and the contaminant of concern (arsenic, nitrate, or lead) is below its maximum contaminant level (arsenic < 10ug/L; nitrate <10mg/L, and lead <15 ug/L)
Well Stewardship Behaviors | 6 and 12 months
  This will be assessed based on questions in the homeowner survey which asks the participants what actions they take to test, treat, and maintain the water quality that is coming from their private well.

SECONDARY OUTCOMES:
Health literacy | 6 months and 12 months
  1. Water Environmental Literacy Level Scale - WELLS is a 6-item scale. The reference for this is: Irvin, V. L., Rohlman, D., Vaughan, A., Amantia, R., Berlin, C., & Kile, M. L. (2019). Development and Validation of an Environmental Health Literacy Assessment Screening Tool for Domestic Well Owners: The Water Environmental Literacy Level Scale (WELLS). International journal of environmental research and public health, 16(5), 881. doi:10.3390/ijerph16050881
  2. Brief Health Literacy Screener (Chew Items) is a 3-item scale. The reference for this: Chew, L.D., Bradley, K.A., & Boyko, E.J. (2004). Brief questions to identify patients with inadequate health literacy. Family Medicine, 36(8): 588-594.
Risk perception | 6 months and 12 months
  This will be assessed our homeowner survey which includes a condensed form of the RANAS (Risk, Attitude, Norms, Ability, Self-Regulation) Scales published in Flannigan et al (2015) Dissemination of well water arsenic results to homeowners in Central Maine: influences on mitigation behavior and continued risks for exposure. Sci Total Environ, 505: 1282-90.

OTHER OUTCOMES:
Health history - Blood pressure | 6 months and 12 months
  National Health and Nutrition Examination Survey (NHANES) questionnaires for Blood Pressure
Health history - Diabetes | 6 months and 12 months
  National Health and Nutrition Examination Survey (NHANES) questionnaires for Diabetes
Health history - Cardiovascular | 6 months and 12 months
  National Health and Nutrition Examination Survey (NHANES) questionnaires for cardiovascular
Health history - Cancer | 6 months and 12 months
  National Health and Nutrition Examination Survey (NHANES) questionnaires for cancer
Health history - Reproductive Health | 6 months and 12 months
  National Health and Nutrition Examination Survey (NHANES) questionnaires for reproductive health
Health history - Anemia | 6 months and 12 months
  National Health and Nutrition Examination Survey (NHANES) questionnaires for anemia
Patient-Reported Quality of life | 6 months and 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale to assess health symptoms (pain, fatigue, mental health, physical health, social health and overall health

CONTACTS AND LOCATIONS:
Overall Officials: Molly Kile, ScD, Principal Investigator — Oregon State University; Veronica Irvin, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Irvin VL, Kile ML, Lucas-Woodruff C, Cude C, Anderson L, Baylog K, Hovell MF, Choun S, Kaplan RM. An overview of the Be Well Home Health Navigator Program to reduce contaminants in well water: Design and methods. Contemp Clin Trials. 2024 May;140:107497. doi: 10.1016/j.cct.2024.107497. Epub 2024 Mar 11. PMID 38471641